CLINICAL TRIAL: NCT07285512
Title: Eating Behaviors in Children and Adolescents With/Without Celiac Disease: A Cross-Sectional and Longitudinal Study
Brief Title: Eating Behaviors in Children and Adolescents With/Without Celiac Disease
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marina Di Stefano, Doctor, IRCCS San Raffaele
Other Study IDs: DAN-CD
Record Dates: First submitted 2025-12-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Celiac Disease in Children; Eating Behaviors
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac disease group: Adolescents aged 11-17 years with a confirmed diagnosis of celiac disease, established according to the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) criteria (positive serology and/or duodenal biopsy). Participants may be at any time point after diagnosis for the cross-sectional component. A sub-cohort diagnosed <6 months prior to enrollment will participate in the longitudinal follow-up at 6, 12, and 24 months. No interventions are administered; participants complete self-report questionnaires (YEDE-Q) and parents complete the PEDE-Q, along with a structured clinical and psychosocial survey.
- Healthy control group: Adolescents aged 11-17 years without celiac disease or other chronic medical conditions requiring dietary therapy. Controls are matched to the CD group by age and sex. They are recruited from the general pediatric population of the hospital and from local schools. Participants complete the same self-report questionnaires (YEDE-Q) and structured survey; parents complete the PEDE-Q. Controls are included only in the cross-sectional comparison.

SUMMARY:
This observational study investigates the prevalence and severity of disordered eating behaviors in adolescents aged 11-17 years with celiac disease. Participants complete validated self-report questionnaires (Youth Eating Disorder Examination Questionnaire, YEDE-Q, and Parent Eating Disorder Examination Questionnaire, PEDE-Q) and a structured clinical form. A healthy control group, matched by age and sex, is included for comparison. A longitudinal sub-cohort diagnosed with celiac disease <6 months prior will be followed at 6, 12, and 24 months to evaluate changes in eating psychopathology and associated clinical variables.

DETAILED DESCRIPTION:
Celiac disease (CD) is a chronic autoimmune condition that requires lifelong adherence to a strict gluten-free diet. Adolescence represents a period of heightened vulnerability for the development of disordered eating behaviors, particularly in chronic conditions requiring dietary restrictions. Emerging evidence suggests that youths with CD may be at increased risk of problematic eating behaviors, including shape and weight concerns, dietary restraint, and loss-of-control eating; however, data in pediatric CD populations are limited and inconsistent.

This study aims to characterize eating-related psychopathology in adolescents aged 11-17 years with a diagnosis of CD, using validated instruments adapted for youth (Youth Eating Disorder Examination Questionnaire, YEDE-Q, and Parent Eating Disorder Examination Questionnaire, PEDE-Q). The study has both a cross-sectional and a longitudinal component.

The cross-sectional component will compare adolescents with CD to age- and sex-matched healthy controls recruited from outpatient pediatric services and local schools. Participants will complete an online self-report questionnaire battery including the YEDE-Q and a structured clinical and psychosocial survey assessing diagnostic history, gastrointestinal symptoms, lifestyle factors, adherence to the gluten-free diet, academic functioning, and co-morbidities. Parents or caregivers will complete the PEDE-Q. The primary outcome is the global score of the YEDE-Q.

The longitudinal component includes a sub-cohort of adolescents diagnosed with CD within the past six months. These participants will be reassessed at 6, 12, and 24 months post-diagnosis to evaluate trajectories of eating psychopathology and identify factors associated with the emergence, persistence, or remission of disordered eating behaviors over time.

No biological samples are collected, and no experimental interventions are administered. All data are obtained through questionnaires. The study is conducted at IRCCS Ospedale San Raffaele, Milan, Italy.

The overarching goal is to improve early recognition of disordered eating in adolescents with CD, inform clinical practice, and contribute foundational data for future preventive interventions in this population.

ELIGIBILITY:
Inclusion Criteria:

Celiac Disease Group (Cases)

* Adolescents aged 11 to 17 years
* Confirmed diagnosis of celiac disease according to the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) criteria (positive serology and/or duodenal biopsy)
* Ability to understand and complete questionnaires in Italian
* For the longitudinal cohort: diagnosis < 6 months prior to enrollment

Healthy Control Group

* Adolescents aged 11 to 17 years
* No diagnosis of celiac disease
* Ability to understand and complete questionnaires in Italian

Exclusion Criteria:

* Significant cognitive impairment or developmental disorders preventing questionnaire completion
* Inadequate understanding of the Italian language
* Refusal or inability to provide assent/consent

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will enroll adolescents aged 11-17 years, including two groups: (1) patients with a confirmed diagnosis of celiac disease, and (2) healthy controls matched by age and sex. Participants in the celiac disease group are recruited from the Pediatric Unit of IRCCS Ospedale San Raffaele and must have a diagnosis established according to ESPGHAN guidelines; a subset diagnosed within the previous 6 months will be included in a longitudinal follow-up. Healthy controls are recruited from outpatient pediatric clinics and local schools and must have no chronic medical conditions requiring dietary therapy. All participants must be able to understand Italian and complete self-report questionnaires, with a caregiver available to complete the parent-report instrument.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Eating Psychopathology - Youth Eating Disorder Examination Questionnaire (YEDE-Q) Global Scores | Baseline (cross-sectional assessment)
  Eating disorder psychopathology will be assessed using the YEDE-Q, completed by the adolescent. This tool evaluates restraint, eating concern, shape concern, and weight concern. The primary endpoint is the global score (range 0-6), with higher values indicating greater eating-related psychopathology.
Eating Psychopathology - Parent Eating Disorder Examination Questionnaire (PEDE-Q) Global Scores | Baseline (cross-sectional assessment)
  Eating disorder psychopathology will be assessed using the PEDE-Q, completed by a caregiver. This tool evaluates restraint, eating concern, shape concern, and weight concern from the point of view of the caregiver. The primary endpoint is the global score (range 0-6), with higher values indicating greater eating-related psychopathology.

SECONDARY OUTCOMES:
Associations Between Eating Psychopathology and Clinical/Psychosocial Variables | baseline
  Associations between YEDE-Q and PEDE-Q global scores and relevant clinical and psychosocial variables will be evaluated. Variables include BMI z-score, diagnostic delay, time since diagnosis, gastrointestinal symptoms, physical activity, adherence to gluten-free diet, school functioning, and medical/psychological comorbidities.
Longitudinal Change in Eating Psychopathology (YEDE-Q Global Score) | 6 months, 12 months, and 24 months after diagnosis
  Among adolescents with a recent diagnosis of celiac disease (<6 months), changes in eating disorder psychopathology over time will be assessed using the Youth Eating Disorder Examination Questionnaire (YEDE-Q). Repeated measures of adolescent-reported global scores (range 0-6) will be collected to evaluate progression, persistence, improvement, or remission of disordered eating symptoms.
Longitudinal Change in Eating Psychopathology (PEDE-Q Global Scores) | 6 months, 12 months, and 24 months after diagnosis
  Among adolescents with a recent diagnosis of celiac disease (<6 months), changes in eating disorder psychopathology over time will be assessed using the Parent Eating Disorder Examination Questionnaire (PEDE-Q). Repeated measures of parent-reported global scores (range 0-6) will be collected to evaluate progression, persistence, improvement, or remission of disordered eating symptoms.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset contains sensitive information from minors regarding health status and eating psychopathology, and sharing identifiable or potentially re-identifiable data is not permitted under institutional and ethical guidelines.